CLINICAL TRIAL: NCT04872205
Title: The Reliability and Validity of the Turkish Version of the Shanghai Elbow Dysfunction Score
Brief Title: The Turkish Version of the Shanghai Elbow Dysfunction Score
Status: Completed | Type: Observational
Sponsor: Istanbul University - Cerrahpasa (Other)
Responsible Party: Principal Investigator, Tansu Birinci, PT, PhD, Istanbul University - Cerrahpasa
Other Study IDs: 33
Record Dates: First submitted 2021-04-30; First posted 2021-05-04 (Actual); Last update posted 2024-10-08 (Actual); Status verified 2024-10

CONDITIONS: Elbow Fracture; Stiffness of Elbow, Not Elsewhere Classified; Orthopedic Disorder; Assessment, Self
Keywords: Elbow; Reliability; Validity; Function; Fracture
MeSH Terms: conditions — Elbow Fractures; Musculoskeletal Diseases; Fractures, Bone

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The Shanghai Elbow Dysfunction Score (SHEDS) is originally developed in English to evaluate elbow function in patients with elbow stiffness. The purpose of this study is to translate and cross-culturally adapt the SHEDS instrument into Turkish and investigate its psychometric properties.

DETAILED DESCRIPTION:
The Shanghai Elbow Dysfunction Score (SHEDS) is originally developed in English to evaluate joint function in patients with elbow stiffness. The purpose of this study is to translate and cross-culturally adapt the SHEDS instrument into Turkish and investigate its psychometric properties. Approximately seventy patients with elbow limitation will be included. For cross-cultural adaptation, two bi-lingual translators will use the back-translation procedure. Within a 3-to-5-day period after the first assessment, the participants will complete the Turkish version of SHEDS (SHEDS-T) to evaluate test-retest reliability. Cronbach's alpha (α) will use to assess internal consistency. The correlation with the Turkish version of the Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire, the Turkish version of Mayo Elbow Performance Score, and Short Form-12 will be determined to check the validity. Responsiveness and floor and ceiling effects will be detected.

ELIGIBILITY:
Inclusion Criteria:

* Aged between 20 and 55 years
* Elbow fracture in the six months before the study
* Elbow limitation in flexion or extension
* Fractures should be managed with surgically
* Being able to follow simple instructions
* Being able to read and write in Turkish

Exclusion Criteria:

* Malunion or Nonunion Fracture
* The occurrence of complex regional pain syndrome, peripheric nerve injury, heterotopic ossification, myositis ossification or post-traumatic ankylosing
* Non-healing wound or infection
* Previously received physiotherapy for elbow limitation
* Having any cardiovascular diseases, neurological disorders, rheumatic diseases or psychiatric diseases
* Shoulder, elbow or wrist movement limitation in contralateral upper extremity or absence of limbs in the contralateral upper extremity

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: All participants are patients who had sustained an elbow fracture and are treated surgically. The participants with elbow stiffness after an elbow fracture are directed for assessment following a confirmation by an orthopaedist that the bone fracture healed based on the physical examinations and diagnostic imaging.
Sampling Method: Non-Probability Sample
Enrollment: 108 (Actual)
Dates: Start 2021-06-30 (Actual); Primary Completion 2021-09-01 (Actual); Study Completion 2022-03-07 (Actual)

PRIMARY OUTCOMES:
The Shanghai Elbow Dysfunction Score (SHEDS) | Baseline (First assessment)
  The Shanghai Elbow Dysfunction Score (SHEDS) is composed of 12 items and developed in 3 parts: elbow motion capacities, elbow-related symptoms, and patient satisfaction level. The SHEDS is a comprehensive and valid scoring system to evaluate elbow function in patients with elbow stiffness.

SECONDARY OUTCOMES:
The Shanghai Elbow Dysfunction Score (SHEDS) | Within a 3-to-5-day period after the first assessment (Second assessment)
  The Shanghai Elbow Dysfunction Score (SHEDS) is composed of 12 items and developed in 3 parts: elbow motion capacities, elbow-related symptoms, and patient satisfaction level. The SHEDS is a comprehensive and valid scoring system to evaluate elbow function in patients with elbow stiffness. The cumulative score is ranged from 0 to 100, where the higher scores indicate an increased level of function.
The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire | Baseline (First assessment)
  The Disabilities of the Arm, Shoulder and Hand (DASH) questionnaire 30 core questions and optional additional 8 questions that are scored on a 5-point Likert-type scale (no difficulty-unable). The cumulative DASH score is ranged from 0 to 100, where the higher scores indicate an increased degree of disability.
Mayo Elbow Performance Score (MEPS) | Baseline (First assessment)
  Mayo Elbow Performance Score (MEPS) is designed to measure pain, stability, range of motion and the patient's ability to accomplish functional tasks, is one of the most commonly used physician based and joint-specific elbow rating system The cumulative MEPS score is ranged from 0 to 100, where the higher scores indicate an increased level of function.
Short Form-12 (SF-12) | Baseline (First assessment)
  Short Form-12 (SF-12), which is developed based on Short Form-36, consists of 12 items: 7 items dealing with the physical components scores (PCS-12) and 5 items related to the mental components scores (MCS-12) of SF-12. Range of both scores is 0 to 100, where the higher scores indicate better health related quality of life.

CONTACTS AND LOCATIONS:
Overall Officials: Tansu Birinci, PhD, Principal Investigator — Istanbul Medeniyet University
Locations (1):
- Istanbul University-Cerrahpasa, Istanbul, Bakırkoy, Turkey (Türkiye)